CLINICAL TRIAL: NCT03961711
Title: Randomized Controlled Trial Assessing Post-operative Telemedicine Versus In-Person Clinic Visits in Hip and Knee Arthroplasty
Brief Title: Telemedicine in Total Hip Arthroplasty and Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hawkins Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00087297
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine encounter (Experimental): Patients will undergo a Telemedicine encounter with the physician at the 3-week post-operative timepoint following a total hip or total knee arthroplasty.
  Interventions: Procedure: Telemedicine
- In-person Clinic Visit (Active Comparator): Patients will undergo an in-person clinic encounter with the physician at the 3-week post-operative timepoint following a total hip or total knee arthroplasty.
  Interventions: Procedure: In-Person Clinic Visit

INTERVENTIONS:
Procedure: Telemedicine — Patients will undergo a Telemedicine encounter with the physician at the 3-week post-operative timepoint following a total hip or total knee arthroplasty.
  Arms: Telemedicine encounter
Procedure: In-Person Clinic Visit — Patients will undergo an in-person clinic encounter with the physician at the 3-week post-operative timepoint following a total hip or total knee arthroplasty.
  Arms: In-person Clinic Visit

SUMMARY:
The objective of this study is to evaluate patient perspective on telemedicine used in 3 week post operative visits for knee and hip arthroplasty. It is hypothesized that patient satisfaction with telemedicine follow-up is equal to patient satisfaction with in-office followup. Patient satisfaction will be assessed at the 3-week and 9-week post-operative timepoints.

DETAILED DESCRIPTION:
In 2014 there were 370,770 total hip replacements and 680,150 total knee replacements performed in the United States. As the elderly proportion of the population continues to grow, it is estimated that the number of total hip arthroplasty will grow by 71 percent and total knee arthroplasty will grow by 85 percent by the year 2030 (Sloan, M The Journal of Bone and Joint Surgery 2018). As these numbers continue to rise, health care delivery must evolve into a more efficient, cost effective system without compromising the quality of the care delivered.

Telemedicine involves using electronic communications and software to provide clinical services to patients in place of an in-person visit. Benefits of telemedicine include avoiding unnecessary trips to hospitals, saving time, and reducing the number of working days missed (Asiri, A Acta Inform Med 2018). Used in general surgery followup care, anonymous survey responses demonstrated a high degree of satisfaction with 85% expressing a desire to utilize telemedicine for followup care in the future (Nikolian, V Annals of Surgery 2018). Postoperative telemedicine has been studied in many specialties, but literature exploring its use in orthopedics has been scant.

ELIGIBILITY:
Inclusion Criteria:

There will be two arms of this study, knee and hip patients.

* Knee: All adult patients over the age of 18 scheduled for a primary total knee arthroplasty will be eligible for the inclusion in the study.
* Hips: All adult patients over the age of 18 scheduled for a primary total hip arthroplasty will be eligible for the inclusion in the study.

Exclusion Criteria:

* lack of access to a telephone
* history of wound complications
* venous thromboembolism (deep vein thrombosis and/or pulmonary embolism),
* significant cardiac history (myocardial infarction, angina, stroke, lower limb ischemia)
* Subject with any condition (including cognitive impairment) that, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Patient reported satisfaction | 9 weeks
  Client Satisfaction Questionnaire (CSQ-8) will be used to assess patient satisfaction of the 3 week encounter both at 3 and 9 weeks post-operatively.
  The scale of the survey ranges from 8-32, with 32 being the best score and 8 being the worst. The higher a patient scores, the more satisfied the patient is with the care provided.

OTHER OUTCOMES:
Patient reported pain level | 9 weeks
  Pain assessed via Visual Analog Score (VAS), 0-10, with 0 being no pain and 10 being extreme pain.
Adverse Events | 9 weeks
  Adverse events will be tracked for both groups and compared.
Time spent during 3-week post-operative encounter | 3 weeks
  Post-operative telemedicine follow up duration compared to clinic follow up duration (measured in minutes).
Patient reported overall quality of life measures | 9 weeks
  Quality of Life assessed via EuroQol-5 Dimensions (EQ-5D) Questionnaire. Levels of perceived problems are coded with 1 being the best outcome and 3 being the worst. The overall health scale portion of the EQ-5D (EQ VAS) is scored on a scale of 0-100, with 100 being the best and 0 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Burnikel, MD, Principal Investigator — Steadman Hawkins Clinic of the Carolinas - Greenville Health System
Locations (1):
- Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No